CLINICAL TRIAL: NCT04442646
Title: Role of "Asthma School" in Disease Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2278CE
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASG= Asthma School Group, with educational intervention (Experimental): experimental "asthma school" group (ASG) will attend control visits as Control Group every three months. In addiction, ASG will attend 3 further meetings consisting in multidisciplinary lessons (pneumologist, nurse, biologist and respiratory therapist) once a week within 1 month after randomization. Study staff will deal with the following topics: asthma physiopathology, recognition of asthma symptoms and exacerbation, educational interventions on therapy and device, nutritional counselling if necessary. Patients will receive a paper diary for symptoms and an expiratory pick flow meter (PFM) to be done twice a day
  Interventions: Behavioral: multidisciplinary lessons
- CG= Control Group, With no educational intervention (No Intervention): Control group will attend control visits every three months.

INTERVENTIONS:
Behavioral: multidisciplinary lessons — the multidisciplinary lessons will be conducted by study staff, formed by pneumologist, nurse, biologist and respiratory therapist once a week within 1 month after randomization. Study staff will deal with the following topics: asthma physiopathology, recognition of asthma symptoms and exacerbation, educational interventions on therapy and device, nutritional counselling if necessary. Patients will receive a paper diary for symptoms and an expiratory pick flow meter (PFM) to be done twice a day
  Arms: ASG= Asthma School Group, with educational intervention

SUMMARY:
According to the definition provided by the GINA guidelines, asthma is characterized by a variable and reversible limitation of expiratory airflow and by the following symptoms: wheezing, dyspnoea, thoracic constriction and/or cough. The type and the severity of airflow limitation can vary over time (1) depending on external agents, such as physical exercise, polluting agents, climate changes and viral infections. The therapy is mainly based on the use of inhaled corticosteroids and bronchodilators. Patients affected by severe asthma (~ 10% of total prevalence of asthma and at high risk of exacerbations and/or hospitalization) may not control their symptoms, even if exposed to maximal doses of inhalation therapy.The behavioural sciences can potentially help to find the psychological factors behind scarce adherence and to develop strategies with the aim of improving the interactive processes between patients, medical doctors and health care professionals

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disease affecting 300 million people worldwide, especially children. In Italy, asthma affects 3 million patients and represents one of the main expenses of the Italian National Heath Care Service. According to the definition provided by the GINA guidelines, asthma is characterized by a variable and reversible limitation of expiratory airflow and by the following symptoms: wheezing, dyspnoea, thoracic constriction and/or cough. The type and the severity of airflow limitation can vary over time (1) depending on external agents, such as physical exercise, polluting agents, climate changes and viral infections. The therapy is mainly based on the use of inhaled corticosteroids and bronchodilators. Patients affected by severe asthma (~ 10% of total prevalence of asthma and at high risk of exacerbations and/or hospitalization) may not control their symptoms, even if exposed to maximal doses of inhalation therapy. More than one third of severe asthma patients receive oral corticosteroids prescriptions, with the risk of severe and irreversible adverse events. Therapy adherence is generally poor when therapeutic regimes are prescribed for chronic diseases, including asthma (4). The behavioural sciences can potentially help to find the psychological factors behind scarce adherence and to develop strategies with the aim of improving the interactive processes between patients, medical doctors and health care professionals (4). Several studies have described intervention models focused on education of the patients to symptoms and exacerbations recognition, therapy management, reduction of the exposure to trigger agents and improvement of social and physical activities (5-6). The intervention is not able to make patients independent in disease managing, but can improve the cooperation in asthma management. Another important aspect in asthma management is the quality of the therapeutic intervention: the correct delivery of inhalation therapy is the key for the disease control (3). Specific educational intervention such as "asthma school" can improve symptoms control and reduce; however, up to day, a universal and standardized protocol is not available and further studies are needed.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosis according to GINA / ATS guidelines.
* Age ≥18 years

Exclusion Criteria:

•cognitive impairment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
number of exacerbations | 2 years
  number of exacerbations in a period of 12 months in asthmatic subjects belonging to experimental group compared to controls.
ER accesses | 2 years
  ER accesses in a period of 12 months in asthmatic subjects belonging to experimental group compared to controls.
number of asthma related hospitalizations | 2 years
  number of asthma related hospitalizations in a period of 12 months in asthmatic subjects belonging to experimental group compared to controls.

SECONDARY OUTCOMES:
Asthma control test ACT (0-25) | 2 years
  evaluating asthma symptoms control in Asthma School Group (ASG) compared to Control Group (CG).
Asthma control questionnaire ACQ (0-6) | 2 years
  evaluating asthma symptoms control in Asthma School Group (ASG) compared to Control Group (CG).
St. George Respiratory questionnaire SGRQ (0-100) | 2 years
  assessing quality of life in Asthma School Group (ASG) compared to Control Group (CG).
airways and systemic inflammation | 2 years
  differential cell count in sputum and blood in Asthma School Group (ASG) compared to Control Group (CG). Sputum inflammatio: number eosinophills >3%, sistemic inflammation: eosiniphils cell count >250 cell/ul
respiratory function | 2 years
  Forced Expiratory Volume in 1 second (FEV1) l, %, Forced Volume Capacity (FVC) l,%, FEV1 / FVC% values in Asthma School Group (ASG) compared to Control Group (CG).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Spanevello, Prof, Principal Investigator — ICS Maugeri
Locations (1):
- Istituti Clinici Maugeri Pneumologia, Tradate, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nair AS, DeMuth K, Chih-Wen Cheng, Wang MD. Asthma Academy: Developing educational technology to improve Asthma medication adherence and intervention efficiency. Annu Int Conf IEEE Eng Med Biol Soc. 2017 Jul;2017:1364-1367. doi: 10.1109/EMBC.2017.8037086. PMID 29060130
- [Background] Klijn SL, Hiligsmann M, Evers SMAA, Roman-Rodriguez M, van der Molen T, van Boven JFM. Effectiveness and success factors of educational inhaler technique interventions in asthma & COPD patients: a systematic review. NPJ Prim Care Respir Med. 2017 Apr 13;27(1):24. doi: 10.1038/s41533-017-0022-1. PMID 28408742
- [Background] Muhlhauser I, Richter B, Kraut D, Weske G, Worth H, Berger M. Evaluation of a structured treatment and teaching programme on asthma. J Intern Med. 1991 Aug;230(2):157-64. doi: 10.1111/j.1365-2796.1991.tb00424.x. PMID 1865168
- [Background] Ringsberg KC, Wiklund I, Wilhelmsen L. Education of adult patients at an "asthma school": effects on quality of life, knowledge and need for nursing. Eur Respir J. 1990 Jan;3(1):33-7. PMID 2311729